CLINICAL TRIAL: NCT00543231
Title: A Pharmacokinetic and Safety Assessment of G3139 Administered by Subcutaneous Injection to Patients With Solid Tumors
Brief Title: A Phase I Study of G3139 Subcutaneous in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GPKS106
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2005-12

CONDITIONS: Tumors
Keywords: ECOG; MRT; NCI CTC; SAE; Short Intravenous Infusion to Patients with Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — oblimersen

INTERVENTIONS:
Drug: G3139, Oblimersen sodium, Bcl-2 antisense oligonucleotide

SUMMARY:
Genasense® is currently administered to subjects in clinical studies as a multiple-day continuous intravenous infusion. Subjects are treated on an outpatient basis and carry a pump that delivers the drug through a peripheral or central intravenous line. The route of administration limits the convenience of treatment, and catheter-related complications have been reported. This study is designed to evaluate the pharmacokinetics and safety of G3139 administered by subcutaneuous injection.

ELIGIBILITY:
Inclusion Criteria:

* A Confirmed diagnosis of a solid tumor malignancy, not to include lymphoma, that has failed standard therapy or for which no standard therapy is available. Patients with a history of brain metastasis will be eligible if there is no evidence of cerebral edema or treatment with steroids.
* Adequate organ function as determined < 7 days prior to starting study medication
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* At least 3 weeks and recovery from effects of major prior surgery or other therapy including radiation therapy, immunotherapy, cytokine, biological, vaccine and chemotherapy

Exclusion Criteria:

* Significant medical diesese
* History of leptomeningeal disease
* Coexisting condition that would require the subject to continue therapy during the treatment phase of the study with a drug known to alter renal function.
* Use of any investigational drug within 3 weeks prior to starting study medication
* Known hypersensitivity to phosphorothioate-containing oligonucleotides
* Pregnancy/Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2005-12; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Institute for Drug Development, San Antonio, Texas, United States